CLINICAL TRIAL: NCT06257394
Title: Multi-center Clinical Trial for Optimal Treatment of Pediatric Very High-risk Acute Lymphoblastic Leukemia in Korea
Brief Title: Treatment of Pediatric Very High-risk Acute Lymphoblastic Leukemia in Korea
Acronym: VHR ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hyoung Jin Kang (Other)
Collaborators: Asan Medical Center (Other); Samsung Medical Center (Other); Severance Hospital (Other); Pusan National University Yangsan Hospital (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Hyoung Jin Kang, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2401-028-1500
Record Dates: First submitted 2024-02-01; First posted 2024-02-14 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-04

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: VHR ALL; NGS-MRD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [Arm A, Dasatinib(Sprycel) Arm] (Experimental): ▪ Arm A : Philadelphia chromosome-positive : Induction (Except Consolidation #3 using Blinatumomab, all administration should be given with Dasatinib.)
  * Morphologic CR after the Induction : Consolidation #1 → Consolidation #2 → Consolidation #3
    1. If MRD & qPCR not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine → DI #1 → IM #2 → DI #2 → Maintenance
    2. If MRD or qPCR positive after the post-consolidation #1 : Consolidation #3 using Blinatumomab →Allogeneic HSCT
  * M2 or M3 after the Induction : Re-induction → Consolidation #2 → Consolidation #3 → Allogeneic HSCT
    1. If MRD & qPCR not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine
    2. If MRD or qPCR positive after the post-reinduction : Consolidation #3 using Blinatumomab
       * In Arm A, except Consolidation #3 using Blinatumomab, all administration should be given with Dasatinib.
  Interventions: Drug: Dasatinib(Sprycel) arm
- [Arm B, Non-Dasatinib(Sprycel) Arm] (Experimental): ▪ Arm B : Other VHR ALL except Philadelphia chromosome-positive : Induction
  * Morphologic CR after the Induction : Consolidation #1 → Consolidation #2 → Consolidation #3
    1. If MRD not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine → Allogeneic HSCT
    2. If MRD positive after the post-consolidation #1 : Consolidation #3 using Blinatumomab →Allogeneic HSCT
  * M2 or M3 after the Induction : Re-induction → Consolidation #2 → Consolidation #3 → Allogeneic HSCT
    1. If MRD not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine
    2. If MRD positive after the post-reinduction : Consolidation #3 using Blinatumomab
  Interventions: Drug: Non-Dasatinib(Sprycel) arm

INTERVENTIONS:
Drug: Dasatinib(Sprycel) arm — ▪ Arm A : Philadelphia chromosome-positive : Induction (Except Consolidation #3 using Blinatumomab, all administration should be given with Dasatinib.)
  * Morphologic CR after the Induction : Consolidation #1 → Consolidation #2 → Consolidation #3
    1. If MRD & qPCR not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine → DI #1 → IM #2 → DI #2 → Maintenance
    2. If MRD or qPCR positive after the post-consolidation #1 : Consolidation #3 using Blinatumomab →Allogeneic HSCT
  * M2 or M3 after the Induction : Re-induction → Consolidation #2 → Consolidation #3 → Allogeneic HSCT
    1. If MRD & qPCR not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine
    2. If MRD or qPCR positive after the post-reinduction : Consolidation #3 using Blinatumomab
       * In Arm A, except Consolidation #3 using Blinatumomab, all administration should be given with Dasatinib.
  Arms: [Arm A, Dasatinib(Sprycel) Arm]
Drug: Non-Dasatinib(Sprycel) arm — ▪ Arm B : Other VHR ALL except Philadelphia chromosome-positive : Induction
  * Morphologic CR after the Induction : Consolidation #1 → Consolidation #2 → Consolidation #3
    1. If MRD not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine → Allogeneic HSCT
    2. If MRD positive after the post-consolidation #1 : Consolidation #3 using Blinatumomab →Allogeneic HSCT
  * M2 or M3 after the Induction : Re-induction → Consolidation #2 → Consolidation #3‡ → Allogeneic HSCT
    1. If MRD not detected after the post-consolidation #1 : Consolidation #3 using HD MTX, HD Cytarabine
    2. If MRD positive after the post-reinduction : Consolidation #3 using Blinatumomab
  Arms: [Arm B, Non-Dasatinib(Sprycel) Arm]

SUMMARY:
Very high-risk acute lymphoblastic leukemia

DETAILED DESCRIPTION:
* Arm A : Philadelphia chromosome-positive : Induction (Except Consolidation #3 using Blinatumomab, all administration should be given with Dasatinib.)

  * Morphologic Complete Remission after the Induction : Consolidation #1 → Consolidation #2 → Consolidation #3

    1. If Minimal Residual Disease & qPCR not detected after the post-consolidation #1 : Consolidation #3 using High Dose Methotrexate, High Dose Cytarabine → DI(Delayed Intensification) #1 → IM(Interim Maintenance) #2 → DI(Delayed Intensification) #2 → Maintenance
    2. If Minimal Residual Disease or qPCR(Quantitative Polymerase Chain Reaction) positivie after the post-consolidation #1 : Consolidation #3 using Blinatumomab →Allogeneic HSCT(Hematopoietic Stem Cell Transplantation)
  * M2 or M3 after the Induction : Re-induction → Consolidation #2 → Consolidation #3 → Allogeneic HSCT(Hematopoietic Stem Cell Transplantation)

    1. If Minimal Residual Disease & qPCR(Quantitative Polymerase Chain Reaction) not detected after the post-consolidation #1 : Consolidation #3 using High Dose Methotrexate, HD Cytarabine
    2. If Minimal Residual Disease or qPCR(Quantitative Polymerase Chain Reaction) positivie after the post-reinduction : Consolidation #3 using Blinatumomab

       * In Arm A, except Consolidation #3 using Blinatumomab, all administration should be given with Dasatinib.
* Arm B : Other VHR ALL except Philadelphia chromosome-positive : Induction

  * Morphologic Complete Remission after the Induction : Consolidation #1 → Consolidation #2 → Consolidation #3

    1. If Minimal Residual Disease not detected after the post-consolidation #1 : Consolidation #3 using High Dose Methotrexate, High Dose Cytarabine → Allogeneic HSCT(Hematopoietic Stem Cell Transplantation)
    2. If Minimal Residual Disease positivie after the post-consolidation #1 : Consolidation #3 using Blinatumomab →Allogeneic HSCT(Hematopoietic Stem Cell Transplantation)
  * M2 or M3 after the Induction : Re-induction → Consolidation #2 → Consolidation #3 → Allogeneic HSCT(Hematopoietic Stem Cell Transplantation)

    1. If Minimal Residual Disease not detected after the post-consolidation #1 : Consolidation #3 using High Dose Methotrexate, High Dose Cytarabine
    2. If Minimal Residual Disease positivie after the post-reinduction : Consolidation #3 using Blinatumomab

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with ALL between the ages of 1 and 19 years at the time of diagnosis who meet one or more of the following conditions:

  * Philadelphia chromosome-positive t(9;22)(q34;q11) or
  * Patients with failed remission who had blast > 5% on bone marrow test after initial remission induction therapy or
  * Hypodiploidy (Number of chromosomes < 44 (less than 44)) or
  * E2A-HLF(Hepatic Leukemia Factor) translocation-positive or
  * When the prognosis is judged to be poor according to NGS-MRD results among high-risk ALL patients (i) In B-ALL, the NGS-MRD(Next Generation Sequencing-Minimal Residual Disease) after consolidation therapy is 0.01% or more, and the NGS-MRD followed during interim maintenance treatment is also 0.01% or more, (ii) In T-ALL, NGS-MRD(Next Generation Sequencing-Minimal Residual Disease) is more than 0.01% after consolidation therapy

Exclusion Criteria:

* Participants with contraindications to medications
* When the study participant or their legal representative withdraws consent
* Pregnant or lactating women (patients of child-bearing potential require adequate contraception during the study period)
* Participants who are medically unsuitable to participate in this study at the discretion of the investigator Participants participating in other interventional studies other than this protocol

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  The time until defined by date of all-cause mortality from the date of 1st infusion
Recurred rate | Up to 5 years
  As the period from enrollment to disease progression/recurrence
Death rate related to infusion | Up to 5 years
  The time until defined by date of drug-related mortality from the date of 1st infusion
Adverse Event | From Day 1 of the clinical trial to 28 days after last drug administration
The rate of Hematopoietic stem cell transplantation | Up to 5 years
  The rate of Hematopoietic stem cell transplantation after the Induction and consolidation therapy

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul saint Mary's Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No